CLINICAL TRIAL: NCT04434092
Title: A Phase III, Randomized, Open-label, Active-controlled, Multicenter Study Evaluating the Efficacy and Safety of Crovalimab Versus Eculizumab in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Not Previously Treated With Complement Inhibitors
Brief Title: A Study Evaluating the Efficacy and Safety of Crovalimab Versus Eculizumab in Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH) Not Previously Treated With Complement Inhibitors
Acronym: COMMODORE 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO42162; 2019-004931-21 (EudraCT Number); 2023-506498-36-00 (EU CTIS Number)
Record Dates: First submitted 2020-06-03; First posted 2020-06-16 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Crovalimab) (Experimental): Crovalimab will be administered at an initial loading dose of 1000 milligrams (mg) (for participants with body weight between 40 and 100 kilograms [kg]) or 1500 mg (for participants with body weight ≥ 100 kg), as intravenous (IV) injection on Day 1 of Week 1 followed by four weekly subcutaneous (SC) injections of 340 mg starting on Day 2 of Week 1 and then once weekly (QW) at Weeks 2,3 and 4. Thereafter crovalimab will be administered, as SC injection, at a maintenance dose of 680 mg (for participants with body weight between 40 and 100 kg) or 1020 mg (for participants with body weight ≥ 100 kg) once every 4 weeks (Q4W) from Week 5 for a total of 24 weeks of study treatment. Participants may continue to receive crovalimab after 24 weeks of treatment up to maximum of 5 years.
  Interventions: Drug: Crovalimab
- Arm B (Eculizumab) (Active Comparator): Participants will receive loading dose of eculizumab 600 mg on Days 1, 8, 15, and 22, followed by maintenance dose of 900 mg on Day 29 and every 2 weeks (Q2W) thereafter until 24 weeks. Participants may switch to receive crovalimab after 24 weeks of eculizumab treatment.
  Interventions: Drug: Crovalimab; Drug: Eculizumab
- Arm C (Crovalimab) (Exploratory) (Experimental): Participants with a body weight ≥ 5 to <12 kg will receive a loading series of crovalimab doses comprised of an IV dose on Day 1 of Week 1, followed by crovalimab SC dose on Day 2 Week 1. Maintenance doses will begin at Week 3 and will be administered Q2W, thereafter. Participants with a body weight ≥ 12 to < 20 kg and ≥ 20 kg will receive a loading series of crovalimab doses comprised of an IV dose on Day 1 of Week 1, followed by weekly crovalimab SC doses for 4 weeks at Week 1 (Day 2) and then at Weeks 2, 3, and 4. Maintenance doses will begin at Week 5 and will be administered Q2W thereafter, for participants with a body weight ≥ 12 to < 20 kg and Q4W thereafter, for participants with a body weight > 20 kg. After 24 weeks of crovalimab treatment, participants who derive benefit from the drug may continue to receive crovalimab.
  Interventions: Drug: Crovalimab

INTERVENTIONS:
Drug: Crovalimab — Dosing depends on body weight. Participants will be dosed as follows:
  * 5 kg to < 12 kg: 100 mg IV on Week 1 Day 1 (W1D1); 85 mg SC on Week 1 Day 2 (W1D2) and Q2W from Week 3 until end of study
  * 12 kg to < 20 kg: 200 mg IV on W1D1; 85 mg SC on W1D2, Weeks 2, 3 and 4; 170 mg SC, Q2W from Week 5 until end of study
  * 20 kg to < 30 kg: 300 mg IV on W1D1; 85 mg SC on W1D2, Weeks 2, 3 and 4; 340 mg SC, Q4W from Week 5 until end of study
  * 30 kg to < 40 kg: 400 mg IV on W1D1; 170 mg SC on W1D2, Weeks 2, 3 and 4; 510 mg SC, Q4W from Week 5 until end of study
  * 40 kg to < 100 kg: 1000 mg IV on W1D1; 340 mg SC W1D2, Weeks 2, 3 and 4; 680 mg SC, Q4W from Week 5 until end of study
  * 100 kg: 1500 mg IV on W1D1; 340 mg SC W1D2, Weeks 2, 3 and 4; 1020 mg SC, Q4W from Week 5 until end of study.
Drug: Eculizumab — Eculizumab will be administered as specified in the respective arm.
  Arms: Arm B (Eculizumab)

SUMMARY:
A study designed to evaluate the non-inferiority of crovalimab compared with eculizumab in participants with PNH who have not been previously treated with complement inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 kg at screening (pediatric participants with body weight < 40 kg)
* Willingness and ability to comply with all study visits and procedures
* Documented diagnosis of PNH, confirmed by high sensitivity flow cytometry
* LDH level ≥ 2x ULN at screening (as per local assessment)
* Vaccination against Neisseria meningitidis serotypes A, C, W, and Y< 3 years prior to initiation of study treatment; or, if not previously done, vaccination administered no later than one week after the first drug administration
* Women of childbearing potential: agreement to remain abstinent or use contraception during the treatment period and for 10.5 months after the final dose of crovalimab or for 3 months after the final dose of eculizumab (or longer if required by the local product label)

Exclusion Criteria:

* Current or previous treatment with a complement inhibitor
* History of allogeneic bone marrow transplantation
* History of Neisseria meningitidis infection within 6 months prior to screening and up to first study drug administration
* History of myelodysplastic syndrome with Revised International Prognostic Scoring System (IPSS-R) prognostic risk categories of intermediate, high and very high
* Pregnant or breastfeeding, or intending to become pregnant during the study, within 10.5 months after the final dose of crovalimab, or 3 months after the final dose of eculizumab (or longer if required by the local product label)
* Participation in another interventional treatment study with an investigational agent or use of any experimental therapy within 28 days of screening or within 5 half-lives of that investigational product, whichever is greater
* Concurrent disease, treatment, procedure or surgery, or abnormality in clinical laboratory tests that could interfere with the conduct of the study, may pose any additional risk for the participant, or would, in the opinion of the Investigator, preclude the participant's safe participation in and completion of the study
* Splenectomy < 6 months before screening
* Positive for Active Hepatitis B and C infection (HBV/HCV)
* History of or ongoing cryoglobulinemia at screening

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2027-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (63):
- Organizacion Medica de Investigacion (OMI), Ciudad Autonoma Buenos Aires, Argentina
- Brazil (3):
  - Centro Integrado de Oncologia de Curitiba, Curitiba, Paraná
  - *X*CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André, São Paulo
  - Beneficencia Portuguesa de Sao Paulo, São Paulo
- China (7):
  - Peking Union Medical College Hospital, Beijing
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Jiangsu Province Hospital, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - Huashan Hospital, Fudan University, Shanghai
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
- France (2):
  - Hopital Claude Huriez - CHU Lille, Lille
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (2):
  - Universitaetsklinkm, Essen
  - Universitaetsklinikum Ulm, Ulm
- General Hospital of Thessaloniki G. Papanikolaou, Thessaloniki, Greece
- Japan (4):
  - Sapporo Medical University Hospital, Hokkaido
  - University of Tsukuba Hospital, Ibaraki
  - NTT Medical Center Tokyo, Tokyo
  - Tokyo Medical University Hospital, Tokyo
- Vilnius University Hospital Santariskiu Clinics, Public Institution, Vilnius, Lithuania
- Malaysia (2):
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Ampang, Ampang, Selangor
- Mexico (2):
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico CITY (federal District)
  - Global Trial Research Center S.A. de C.V., Monterrey, Nuevo León
- Amsterdam UMC, Locatie AMC, Amsterdam, Netherlands
- Philippines (3):
  - Mary Mediatrix Medical Center, Lipa City
  - Philippine General Hospital, Manila
  - St Lukes Medical Center, Quezon
- Poland (5):
  - Szpital Uniwersytecki nr2 im. dr J. Biziela, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Lublin
  - Pratia Poznan, Skórzewo
  - MTZ Clinical Research Powered by Pratia, Warsaw
- Portugal (3):
  - Centro Hospitalar do Baixo Vouga E.P.E. - Hospital de Aveiro, Aveiro
  - Instituto Portugues Oncologia de Lisboa Francisco Gentil EPE, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
- Romania (2):
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Hospital de Basurto, Bilbao, Albacete
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
- Taiwan (2):
  - Chang Gung Medical Foundation - Kaohsiung, Kaohisung
  - National Taiwan Universtiy Hospital, Taipei
- Thailand (3):
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - King Chulalongkorn Memorial Hospital, Pathum Wan
- Ondokuz Mayis Univ. Med. Fac., Samsun, Turkey (Türkiye)
- Medical Center OK!Clinic+, Kyiv, KIEV Governorate, Ukraine
- United Kingdom (2):
  - St James University Hospital, Leeds
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Kulasekararaj AG, Nishimura JI, Roth A, Beveridge L, Buatois S, Buri M, Compagno N, Luder Y, Sreckovic S, Scheinberg P. Managing transient immune complex reactions in patients with paroxysmal nocturnal hemoglobinuria: clinical observations from the COMMODORE 1 and 2 studies. Ther Adv Hematol. 2025 Sep 17;16:20406207251359246. doi: 10.1177/20406207251359246. eCollection 2025. PMID 40978458
- [Derived] Roth A, Fu R, He G, Alzahrani H, Chou SC, Hicheri Y, Kazmierczak M, Recova VL, Uchiyama M, Vladareanu AM, Beveridge L, Buatois S, Buri M, Compagno N, Shi D, Balachandran N, Sreckovic S, Scheinberg P. Safety of Crovalimab Versus Eculizumab in Patients With Paroxysmal Nocturnal Haemoglobinuria (PNH): Pooled Results From the Phase 3 COMMODORE Studies. Eur J Haematol. 2025 Feb;114(2):373-382. doi: 10.1111/ejh.14339. Epub 2024 Nov 13. PMID 39535306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at centres in Argentina, Brazil, China, France, Greece, Germany, Hong Kong, Japan, Lithuania, Malaysia, Mexico, Netherlands, Philippines, Poland, Portugal, Romania Republic of Korea, Singapore, Spain, Sweden, Thailand, Türkiye, Taiwan, Ukraine, and United Kingdom from 08 Oct 2020 to 16 Nov 2022. The study is ongoing.
Pre-assignment Details: A total of 204 participants who were diagnosed with paroxysmal nocturnal hemoglobinuria (PNH) and who had not been previously treated with a complement-inhibitor therapy were randomized in a ratio of 2:1, 135 to crovalimab (Arm A) and 69 to eculizumab (Arm B). 6 paediatric participants were enrolled into non-randomized crovalimab (Arm C).
Groups:
- Arm A: Crovalimab: Crovalimab was administered at an initial loading dose of 1000 milligram (mg) (for participants with body weight between 40 and 100 kilogram (kg)) or 1500 mg (for participants with body weight >=100kg), as intravenous (IV) injection on Day 1 of Week 1 followed by four weekly subcutaneous (SC) injections of 340 mg starting on Day 2 of Week 1 and then once weekly (QW) at Weeks 2,3 and 4. Thereafter crovalimab was administered, as SC injection, at a maintenance dose of 680 mg (for participants with body weight between 40 and 100kg) or 1020 mg (for participants with body weight >=100kg) once every 4 weeks (Q4W) from Week 5 until 24 weeks in primary treatment period. After Week 24, participants continued to receive maintenance dose of crovalimab up to a maximum of 5 years in the extension treatment period.
- Arm B: Eculizumab: Participants received loading doses of eculizumab 600 mg IV on Days 1, 8, 15, and 22, followed by maintenance doses of 900 mg IV on Day 29 and every 2 weeks (Q2W) thereafter up to Week 24 in the primary treatment period. Participants who switched to crovalimab received crovalimab as an IV loading dose of 1000 mg (if body weight was between 40 kg to <100 kg) or 1500 mg (if body weight was >=100kg) on Week 25 Day 1, 340 mg SC on Week 25 Day 2, then 340 mg SC QW on Weeks 26, 27, 28, followed by crovalimab maintenance dose of 680 mg SC (if body weight was between 40 kg to <100 kg) or 1020 mg SC (if body weight was >=100kg) on Week 29 and Q4W thereafter up to a maximum of 5 years in the extension treatment period.
- Arm C: Crovalimab: Pediatric participants received initial loading dose of 1000 mg (for participants with body weight between 40 and 100 kg) or 1500 mg (for participants with body weight >=100kg), as IV injection on Day 1 of Week 1 followed by four weekly SC injections of 340 mg starting on Day 2 of Week 1 and then QW at Weeks 2,3 and 4. Thereafter crovalimab was administered, as SC injection, at a maintenance dose of 680 mg (for participants with body weight between 40 and 100kg) or 1020 mg (for participants with body weight >=100kg) Q4W from Week 5 until 24 weeks in primary treatment period. After Week 24, participants continued to receive maintenance dose of crovalimab up to a maximum of 5 years in the extension treatment period.
Period: Primary Treatment Period:Baseline-Week24
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab | Arm C: Crovalimab
Started | 135 | 69 | 6
Completed | 129 | 68 | 6
Not Completed | 6 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 1 | 1 | 0
Period: Extension Treatment Period:Week 25-5 Yrs
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab | Arm C: Crovalimab
Started | 129 | 68 | 6
Completed | 0 | 0 | 0
Not Completed | 129 | 68 | 6
Not completed — Treatment (Crovalimab) Ongoing | 127 | 65 | 6
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Participant Population includes all participant enrolled to the originally assigned treatment arms (Arms A, B and C).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab | Arm C: Crovalimab | Total
Number analyzed (Participants) | 135 | 69 | 6 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 6 | 8
  Between 18 and 65 years | 122 | 58 | 0 | 180
  >=65 years | 13 | 9 | 0 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 34 | 2 | 94
  Male | 77 | 35 | 4 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 6 | 1 | 25
  Not Hispanic or Latino | 114 | 61 | 5 | 180
  Unknown or Not Reported | 3 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 86 | 51 | 5 | 142
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 4
  White | 45 | 16 | 0 | 61
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Transfusion Avoidance (TA)
Description: TA is defined as participants who are packed red blood cell (pRBC) transfusion-free and do not require transfusion per protocol-specified guidelines. 95% Confidence Interval (CI) for percentage of participants with TA was calculated using the Wilson's method with continuity correction. Participants who withdrew before Week 25 were deemed to have had a transfusion. Percentages are rounded off to the nearest single decimal.
Time Frame: Baseline to Week 25
Population: Primary Analysis Population (PAP) included all randomized participants in Arms A and B who received at least one dose of the originally assigned treatment and having at least one valid lactate dehydrogenase (LDH) level assessment by the central laboratory after the first IV infusion by planned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab
Number analyzed (Participants) | 134 | 69
percentage of participants | 65.7 [56.91 to 73.52] | 68.1 [55.67 to 78.53]
Statistical Analysis 1: Comparison: Arm A: Crovalimab vs Arm B: Eculizumab; Test type: Non-Inferiority — Non-inferiority is met when the lower limit of the 95% CI is greater than -20%; Weighted Difference in Proportion = -2.8, 95% CI 2-sided [-15.67 to 11.14] — 95% CI for the difference in proportions of participants with TA is calculated by Stratified Newcombe CI method

2. Primary Outcome: Percentage of Participants With Hemolysis Control Measured by LDH
Description: A Generalized Estimating Equation (GEE) was used to estimate the population-average percentage of the participants with hemolysis control (measured by LDH ≤1.5 x upper limit of normal (ULN)) from Week 5 to Week 25 taking account of the intra-patient and inter-patient correlation between LDH control statuses across visits. Percentages are rounded off to the nearest single decimal.
Time Frame: Week 5 to Week 25
Population: PAP included all randomized participants in Arms A and B who received at least one dose of the originally assigned treatment and having at least one valid LDH level assessment by the central laboratory after the first IV infusion by planned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab
Number analyzed (Participants) | 134 | 69
percentage of participants | 79.3 [72.86 to 84.48] | 79.0 [69.66 to 85.99]
Statistical Analysis 1: Comparison: Arm A: Crovalimab vs Arm B: Eculizumab; Test type: Non-Inferiority — Non-inferiority is met if the lower limit of the 95% confidence interval (CI) for the odds ratio is above 0.2; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.57 to 1.82]

3. Secondary Outcome: Percentage of Participants With Breakthrough Hemolysis (BTH)
Description: BTH was defined as at least one new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, shortness of breath [dyspnea], anemia [hemoglobin < 10 grams per deciliter (g/dL)], major adverse vascular event [MAVE, including thrombosis], dysphagia, or erectile dysfunction) in the presence of elevated LDH ≥2xULN after a prior LDH reduction to ≤1.5xULN from the start of study treatment. 95% CI for percentage of participants with BTH was calculated using the Wilson's method with continuity correction. Participants who withdrew before Week 25 were deemed to have experienced a BTH event. Percentages are rounded off to the nearest single decimal.
Time Frame: Baseline to Week 25
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab
Number analyzed (Participants) | 134 | 69
percentage of participants | 10.4 [6.04 to 17.21] | 14.5 [7.54 to 25.50]
Statistical Analysis 1: Comparison: Arm A: Crovalimab vs Arm B: Eculizumab; Test type: Non-Inferiority — Non-inferiority is met if the upper limit (UL) of the 95% CI for the difference between crovalimab and eculizumab in the proportion of participants with BTH is less than the non-inferiority margin of 20%; Weighted Difference in Proportion = -3.9, 95% CI 2-sided [-14.82 to 5.26] — 95% CI for the difference in proportions of participants is calculated by Stratified Newcombe CI method

4. Secondary Outcome: Percentage of Participants With Stabilization of Hemoglobin
Description: Stabilized hemoglobin is defined as avoidance of a >= 2 g/dL decrease in hemoglobin level from baseline, in the absence of transfusion. 95% CI for percentage of participants with stabilized hemoglobin was calculated using the Wilson's method with continuity correction. Participants who withdrew before Week 25 were deemed to not have had hemoglobin stabilization. Percentages are rounded off to the nearest single decimal.
Time Frame: Baseline to Week 25
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab
Number analyzed (Participants) | 134 | 69
percentage of participants | 63.4 [54.63 to 71.45] | 60.9 [48.35 to 72.17]
Statistical Analysis 1: Comparison: Arm A: Crovalimab vs Arm B: Eculizumab; Test type: Non-Inferiority — Non-inferiority is met when the lower limit of the 95% CI is greater than -20%; Weighted Difference in Proportion = 2.2, 95% CI 2-sided [-11.37 to 16.31] — 95% CI for the difference in proportions of participants is calculated by Stratified Newcombe CI method

5. Secondary Outcome: Change From Baseline in Fatigue Assessed by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale
Description: Fatigue was assessed using FACIT-F scale. FACIT-F is a self-assessment questionnaire with a 7-day recall period and 13 items evaluating fatigue and its impact on daily life activities. Items are scored on a response scale that ranges from 0 ("not at all") to 4 ("very much so"). Relevant items are reverse scored, and all the items are summed to create a total score range from 0 to 52, with 0 being the worst possible score and 52 being the best possible score. A higher score indicates low fatigue severity. A positive mean change indicates improvement. FACIT-F was assessed in adult participants only.
Time Frame: Baseline to Week 25
Population: PAP included all randomized participants in Arms A and B who received at least one dose of the originally assigned treatment and having at least one valid LDH level assessment by the central laboratory after the first IV infusion by planned treatment. Overall number of participants analyzed is the number of participants ≥18 years with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab
Number analyzed (Participants) | 134 | 67
score on scale
  Baseline | 36.02 (0.877) | 35.09 (1.408)
  Change at Week 25: number analyzed (Participants) | 128 | 66
  Change at Week 25 | 7.79 (0.661) | 5.15 (0.880)
Statistical Analysis 1: Comparison: Arm A: Crovalimab vs Arm B: Eculizumab; Test type: Non-Inferiority — The non-inferiority margin was a -5 point score, where higher scores indicated less fatigue, and hence non-inferiority hypothesis was tested comparing the lower limit of the 95% CI for the difference with a non-inferiority margin of -5 points; Difference in Adjusted mean = 2.64, 95% CI 2-sided [0.68 to 4.60], Standard Error of Mean 0.993 — Non-inferiority is met when the lower limit of the 95% CI is greater than -5

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs are reported based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0.
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2028-09

7. Secondary Outcome: Percentage of Participants With Injection-Site Reactions, Infusion-Related Reactions, Hypersensitivity and Infections (Including Meningococcal Meningitis)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. Injection-site reactions or infusion-related reaction are AEs related to the injection site that occur during or within 24 hours after study drug administration that are judged to be related to the study drug injection.
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2028-09

8. Secondary Outcome: Percentage of Participants With AEs Leading to Study Drug Discontinuation
Description: as for outcome 6
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2028-09

9. Secondary Outcome: Percentage of Participants With Clinical Manifestations of Drug-Target-Drug Complex (DTDC) Formation Amongst Participants Who Switched to Crovalimab Treatment From Eculizumab Treatment
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2028-09

10. Secondary Outcome: Serum Concentrations of Crovalimab And Eculizumab Over Time
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2028-09

11. Secondary Outcome: Percentage of Participants With Anti-Crovalimab Antibodies
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2028-09

12. Secondary Outcome: Change in Pharmacodynamic (PD) Biomarkers Including Complement Activity (CH50) Over Time
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2028-09

13. Secondary Outcome: Change Over Time in Free C5 Concentration in Crovalimab-Treated Participants
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2028-09

14. Secondary Outcome: Observed Value in Reticulocyte Count (Count/Milliliters [mL])
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2028-09

15. Secondary Outcome: Observed Value in Haptoglobin (Milligrams Per Deciliter [mg/dL])
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2028-09

16. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count
Time Frame: Baseline, Day 1 Week 1, Week 2, 3, 4, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23 and 25
Population: Randomized Safety Population includes all randomized participants who have received at least one dose of study treatment. Includes only participants from Arms A and B. Overall number of participants analyzed is the number of participants ≥18 years with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter (L)
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab
Number analyzed (Participants) | 79 | 35
10^9 cells/liter (L)
  Baseline | 2865.56 (22637.24) | 164.26 (114.27)
  Change at Week 1 Day 1: number analyzed (Participants) | 1 | 0
  Change at Week 1 Day 1 | -58.50 (NA) — The standard deviation was not estimable due to low number of participants |
  Change at Week 2: number analyzed (Participants) | 64 | 31
  Change at Week 2 | 542.90 (4314.07) | 105.88 (601.77)
  Change at Week 3: number analyzed (Participants) | 66 | 29
  Change at Week 3 | -71.08 (533.01) | -15.62 (53.79)
  Change at Week 4: number analyzed (Participants) | 63 | 30
  Change at Week 4 | 8.52 (58.01) | -10.56 (51.36)
  Change at Week 5: number analyzed (Participants) | 64 | 30
  Change at Week 5 | -1126.63 (9074.19) | 4.85 (49.43)
  Change at Week 7: number analyzed (Participants) | 57 | 30
  Change at Week 7 | -3517.66 (26606.21) | 7020.33 (38344.72)
  Change at Week 9: number analyzed (Participants) | 63 | 29
  Change at Week 9 | 12.60 (62.05) | 20.65 (60.04)
  Change at Week 11: number analyzed (Participants) | 67 | 28
  Change at Week 11 | 425.66 (3343.99) | 26.12 (81.80)
  Change at Week 13: number analyzed (Participants) | 62 | 28
  Change at Week 13 | 24.47 (48.92) | 28.61 (78.48)
  Change at Week 15: number analyzed (Participants) | 63 | 30
  Change at Week 15 | -838.52 (6735.13) | 37.20 (77.52)
  Change at Week 17: number analyzed (Participants) | 66 | 30
  Change at Week 17 | 1929.82 (15576.37) | 33.22 (73.34)
  Change at Week 19: number analyzed (Participants) | 65 | 30
  Change at Week 19 | 62.91 (390.39) | 22.16 (70.68)
  Change at Week 21: number analyzed (Participants) | 64 | 30
  Change at Week 21 | 633.95 (4919.97) | 15.90 (72.72)
  Change at Week 23: number analyzed (Participants) | 63 | 31
  Change at Week 23 | 698.79 (5409.05) | 27.51 (85.87)
  Change at Week 25: number analyzed (Participants) | 71 | 33
  Change at Week 25 | 1396.46 (11622.57) | 32.31 (97.79)

17. Secondary Outcome: Change From Baseline in Free Hemoglobin
Time Frame: Baseline, Week 2, 3, 4, 5, 9, 13, 17, 21, and 25
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: milligram per litre (mg)/L
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab
Number analyzed (Participants) | 84 | 42
milligram per litre (mg)/L
  Baseline | 474.88 (276.49) | 495.69 (393.56)
  Change at Week 2: number analyzed (Participants) | 79 | 41
  Change at Week 2 | -406.39 (273.33) | -407.10 (339.84)
  Change at Week 3: number analyzed (Participants) | 78 | 40
  Change at Week 3 | -409.10 (286.35) | -393.20 (352.22)
  Change at Week 4: number analyzed (Participants) | 79 | 41
  Change at Week 4 | -413.16 (281.40) | -418.00 (441.01)
  Change at Week 5: number analyzed (Participants) | 77 | 42
  Change at Week 5 | -386.62 (424.67) | -421.14 (402.64)
  Change at Week 9: number analyzed (Participants) | 78 | 41
  Change at Week 9 | -404.29 (298.64) | -405.89 (425.73)
  Change at Week 13: number analyzed (Participants) | 79 | 40
  Change at Week 13 | -409.94 (298.14) | -328.56 (586.25)
  Change at Week 17: number analyzed (Participants) | 78 | 41
  Change at Week 17 | -408.15 (285.24) | -340.00 (503.24)
  Change at Week 21: number analyzed (Participants) | 77 | 40
  Change at Week 21 | -367.86 (341.53) | -387.63 (462.10)
  Change at Week 25: number analyzed (Participants) | 77 | 38
  Change at Week 25 | -431.50 (277.83) | -334.96 (516.40)

18. Secondary Outcome: Change From Baseline in Haptoglobin
Time Frame: Baseline, Week 2, 3, 4, 5, 9, 13, 15, 17, 21, and 25
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: gram (g)/L
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab
Number analyzed (Participants) | 85 | 42
gram (g)/L
  Baseline | 0.05 (0.00) | 0.05 (0.00)
  Change at Week 2: number analyzed (Participants) | 81 | 41
  Change at Week 2 | 0.05 (0.14) | 0.08 (0.19)
  Change at Week 3: number analyzed (Participants) | 80 | 41
  Change at Week 3 | 0.05 (0.16) | 0.11 (0.28)
  Change at Week 4: number analyzed (Participants) | 80 | 41
  Change at Week 4 | 0.08 (0.21) | 0.12 (0.28)
  Change at Week 5: number analyzed (Participants) | 78 | 42
  Change at Week 5 | 0.06 (0.16) | 0.09 (0.23)
  Change at Week 9: number analyzed (Participants) | 78 | 41
  Change at Week 9 | 0.05 (0.17) | 0.07 (0.23)
  Change at Week 13: number analyzed (Participants) | 80 | 39
  Change at Week 13 | 0.04 (0.17) | 0.06 (0.21)
  Change at Week 17: number analyzed (Participants) | 78 | 41
  Change at Week 17 | 0.05 (0.16) | 0.05 (0.14)
  Change at Week 21: number analyzed (Participants) | 78 | 40
  Change at Week 21 | 0.06 (0.18) | 0.06 (0.22)
  Change at Week 25: number analyzed (Participants) | 77 | 39
  Change at Week 25 | 0.06 (0.17) | 0.05 (0.21)

ADVERSE EVENTS:
Time Frame: From randomization until primary completion date cutoff (up to approximately 25 weeks) Data collected up to 25 weeks are reported here. Adverse event data collection for the Extension Treatment Period is ongoing and will be reported one year after the study completion date.
Description: All Participant Population includes all participant enrolled to the originally assigned treatment arms (Arms A, B and C).
Arm/Group | Arm A: Crovalimab | Arm B: Eculizumab | Arm C: Crovalimab
All-Cause Mortality (participants affected / at risk) | 2/135 | 1/69 | 0/6
Serious Adverse Events (participants affected / at risk) | 22/135 | 14/69 | 0/6
Other Adverse Events (participants affected / at risk) | 102/135 | 55/69 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Crovalimab (N=135) | Arm B: Eculizumab (N=69) | Arm C: Crovalimab (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 2 (4) | 1 (1) | 0 (0)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Central nervous system infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Crovalimab (N=135) | Arm B: Eculizumab (N=69) | Arm C: Crovalimab (N=6)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 15 (18) | 8 (11) | 1 (1)
Type III immune complex mediated reaction (Immune system disorders) | 0 (0) | 11 (12) | 0 (0)
COVID-19 (Infections and infestations) | 28 (28) | 9 (9) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 17 (21) | 11 (14) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (8) | 5 (5) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 20 (21) | 10 (12) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 7 (7) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 18 (45) | 8 (15) | 0 (0)
White blood cell count decreased (Investigations) | 17 (46) | 10 (29) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 11 (17) | 7 (17) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (12) | 7 (16) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (34) | 9 (25) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (8) | 1 (2) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 4 (13) | 0 (0)
Headache (Nervous system disorders) | 13 (17) | 6 (9) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT04434092/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT04434092/SAP_001.pdf